CLINICAL TRIAL: NCT06182735
Title: A Phase I Clinical Study to Assess the Safety and Efficacy of CD70-targeted CAR-NKT in the Treatment of Relapsed or Metastatic Advanced Renal Cell Carcinoma.
Brief Title: CD70-targeted CAR-NKT Cells(CGC729) Therapy in the Renal Cell Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Head of Urology Department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGC729-IIT-01
Record Dates: First submitted 2023-12-06; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyclophosphamide + Fludarabine + Infusion of CAR-NKT Cells (Experimental): Lymphodepleting regimen, Cyclophosphamide 250mg/m2 IV on day -5 to -3 and Fludarabine 25mg/m2 IV on days -5 to -3. Followed by infusion of CAR-NKT on day 0.
  Potential CGC729 doses:
  Dose level 1: 5.0×106 CAR- NKT cells/m2; Dose level 2: 1.5×107 CAR- NKT cells/m2; Dose level 3: 4.5×107 CAR- NKT cells/m2.
  Interventions: Combination Product: Cyclophosphamide + Fludarabine + Infusion of CAR-NKT Cells

INTERVENTIONS:
Combination Product: Cyclophosphamide + Fludarabine + Infusion of CAR-NKT Cells — Biological: CD70 CAR-NKT cells. Drug: Cyclophosphamide. Drug: Fludarabine.

SUMMARY:
This is a phase I, open-label, single-arm study conducted to evaluate the safety, tolerability, PK, and preliminary efficacy of CGC729 with Relapsed or Metastatic advanced renal cell carcinoma.

Condition or disease:Renal Cell Carcinoma Intervention/treatment: Biological: CD70 CAR-NKT cells Phase 1

DETAILED DESCRIPTION:
Dose exploration for this study will be a 3+3 design with a target DLT rate of <1/3. A particular dose level will be expanded to 6 patients if one patient out of 3 patients treated at that particular dose level develops DLT. Once this occurs, further dose-escalations are halted until the dose has proven to be safe in the expanded cohort. If 2 or more in a cohort of 6 patients develop DLT no further dose escalation is allowed, and the next lower dose level will be expanded to 6 patients in total. The highest dose among the dose levels tested at which no more than one out of six patients experiences DLT will be considered the MTD. Dose exploration can be discontinued once one or more dose levels with an acceptable safety profile and satisfactory antitumor activity have been selected for subsequent evaluation.

During the treatment period of the study, three dose levels of CGC729 will be evaluated. Each of the dose levels will evaluate the safety of the CAR-NKT cells.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects or their guardians agree to participate in this clinical trial and sign the ICF, indicating that they understand the purpose and procedures of this clinical trial and are willing to participate in the research.
2. Age 18 to 75 years.
3. Patients with advanced clear cell renal cell carcinoma confirmed by histology or cytology to be recurrent or metastatic after at least second-line treatment.
4. Archival and/or fresh tumor tissue samples are required.
5. At least one measurable lesion at baseline per RECIST version 1.1.
6. ECOG 0-1 points.
7. The expected survival time is more than 12 weeks.
8. The functions of important organs are basically normal: Hematopoietic function: neutrophils 1.5×109/L, platelets 75×109/L, hemoglobin 80g/L; Renal function: creatinine clearance of ≥60 mL/min.; Liver function: ALT and AST≤2.5×ULN (≤5 × ULN for patients with liver metastases); Total bilirubin≤1.5×ULN. Coagulation INR < 1.7.
9. Pregnancy tests for women of childbearing age shall be negative, Both men and women agreed to use effective contraception.

Exclusion Criteria:

1. Pregnant or lactating female subjects.
2. Pregnant or lactating female subjects.
3. Known positive test result for human immunodeficiency virus (HIV) oracquired immune deficiency syndrome (AIDS).
4. Active infection or uncontrollable infection.
5. Known to have active or uncontrolled autoimmune diseases, such as Crohns disease, rheumatoid arthritis, systemic lupus erythematosus, etc. .
6. Having a history of any mental illness, including dementia, altered mental status, which may affect informed consent and the understanding of the subject by the relevant questionnaire.
7. Have a serious uncontrollable illness that may affect the subject receiving treatment for this study.
8. Subjects with other malignant tumors within the past 2 years, except basal or squamous skin cancer, superficial bladder cancer, and breast cancer in situ, have been completely cured and do not need follow-up treatment.
9. Subjects who are using systemic steroids or steroid inhalers for treatment.
10. Use of anti-CD70 therapy or cell therapy within the previous 3 months.
11. Immunotherapy, targeted drug therapy or chemotherapy within 5 drug half-lives within 2 weeks before cell infusion.
12. Subjects allergic to immunotherapy or related drugs.
13. Patients with leptomeningeal metastasis or central nervous system metastasis, and definite central nervous system underlying diseases with significant symptoms in the past 6 months.
14. Subjects with NYHA heart failure class ≥2 or hypertension uncontrolled by standard therapy requiring special treatment, previous history of myocarditis, or myocardial infarction within 6 months.
15. Earnestly received or organ transplantation or preparing to receive organ transplants.
16. Other investigators deem it unsuitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-01-28 (Estimated); Study Completion 2025-01-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing DLT | Day 28 after CGC729 infusion
  1.Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs) Dose limiting toxicity (DLT) is an AE that meets the following criteria and occurs within 28 days of CGC729 infusion.AE is graded according to CTCAE version 5.0.

SECONDARY OUTCOMES:
ORR of CD70 CAR-NKT cell dynamics. | Day 1 through week 52
  Assess Objective response rate(ORR)
DCR of CD70 CAR-NKT cell dynamics. | Day 1 through week 52
  Disease control rate (DCR)
The safey of CD70 CAR-NKT cell dynamics | Day 1 through week 52
  Adverse events (AEs) of CD70 CAR-NKT cell dynamics, Duration and severity of AEs,AE is graded according to CTCAE version 5.0.
Cmax of CD70 CAR-NKT cell dynamics. | Day 1 through week 52
  Peak Plasma Concentration
Tmax of CD70 CAR-NKT cell dynamics. | Day 1 through week 52
  Time to Maximum Plasma Concentration
AUC of CD70 CAR-NKT cell dynamics. | Day 1 through week 52
  Area under the plasma concentration versus time curve

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Principal Investigator — Fudan University; Dingwei Ye, Principal Investigator — Fudan University
Locations (1):
- Jian Zhang, Shanghai, China

IPD SHARING:
Plan to Share IPD: No